CLINICAL TRIAL: NCT02034162
Title: A Double-Blind, Randomized, Multi-Center, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a Single Dose of a 500-mg Chewable Tablet of Mebendazole in the Treatment of Soil-Transmitted Helminth Infections (Ascaris Lumbricoides and Trichuris Trichiura) in Pediatric Subjects
Brief Title: A Study to Assess the Efficacy and Safety of Mebendazole for the Treatment of Helminth Infections in Pediatric Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100933; MEBENDAZOLGAI3003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Helminth Infections
Keywords: Helminth infections; Helminths; Pediatric; Preschool aged; School aged; Mebendazole; Vermox; Placebo
MeSH Terms: conditions — Trematode Infections | interventions — Mebendazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mebendazole (Active Comparator): Mebendazole will be administered as a single 500-mg chewable tablet in a double-blind manner at the baseline visit (Day 1) and in an open-label manner at Visit 4 (Day 21).
  Interventions: Drug: Mebendazole
- Placebo (Placebo Comparator): Matching placebo will be administered as a single-dose chewable tablet in a double-blind manner at the baseline visit (Day 1).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mebendazole — Mebendazole will be administered as a single-dose 500 mg chewable tablet. For children 1 year to <36 months of age, the tablet will be placed in a teaspoon and bottled water will be poured into the remaining volume of the teaspoon. The tablet will then be allowed to absorb all water (absorption time has been observed to take less than 1 minute) to become a soft semi-solid mass without any hard particles. This semi-solid form can then be easily ingested by the child.
  Arms: Mebendazole
Drug: Placebo — Matching placebo will be administered as a single-dose chewable tablet. For children 1 year to <36 months of age, the tablet will be placed in a teaspoon and bottled water will be poured into the remaining volume of the teaspoon. The tablet will then be allowed to absorb all water (absorption time has been observed to take less than 1 minute) to become a soft semi-solid mass without any hard particles. This semi-solid form can then be easily ingested by the child.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mebendazole compared with placebo in pediatric participants with Helminth infections.

DETAILED DESCRIPTION:
This will be a double-blind (neither physician nor participant knows the treatment that the participant receives), randomized (the study drug is assigned by chance), multi-center, parallel-group study (each group of participants will be treated at the same time) to evaluate the efficacy and safety of mebendazole (a drug currently being investigated for Helminth gastrointestinal infections) compared with placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial) in children (including pre-school and school-aged children) with Helminth infections. The study will consist of 3 phases: a screening phase, a double-blind treatment phase, and a post-treatment (or follow-up) phase. A pharmacokinetic (explores what a drug does to the body) open-label substudy (asks a separate research question from the parent study while using the same participant population but does not contribute to the parent study's objectives) will be included in the parent study to measure the level of mebendazole in the blood. Safety assessments will be performed throughout the study. Each participant will take part in the study for approximately 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are >=9 years old must have a negative urine pregnancy test at screening or at the time of randomization
* Participants must be an otherwise healthy child, based on medical history, physical examination, vital signs, hemoglobin, and concomitant medications
* Participants >=3 years of age must have teeth and be able to chew
* Participant must be available to return to the study site for all visits, including the follow-up visit
* Parent(s)/guardians of participants (or their legally-accepted representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to have their child participate in the study
* Children 6 years of age and older will be asked to assent (agree) to their participation using appropriate language to their level of understanding; assent will be documented

Exclusion Criteria:

* Participant has active diarrhea (defined as the passage of 3 or more loose or liquid stools per day) at screening or at the time of randomization
* Participant has a significant medical disorder, participant has difficulty in chewing or swallowing
* Participant has significant anemia (<8 g/dL)
* Participant has significant wasting (greater than 2 standard deviations below the mean World Health Organization [WHO] Child Growth Standards for weight-for-height or body mass index)
* Participant has a known hypersensitivity to mebendazole, any inert ingredients in the chewable formulation
* Participant has preplanned surgery/procedures that would interfere with the conduct of the study during the course of study
* Participants has received an investigational drug (including vaccines) or used an investigational medical device within 30 days before the planned start of treatment, or is currently enrolled in an investigational study
* Employees of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator
* Participant has taken any form of medication containing mebendazole or any other treatment for soil transmitted helminth infection within 30 days of entry into the study

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Ethiopia (2):
  - Gonder
  - Jimma
- Kigali, Rwanda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 8-Dec-2014 to 3-Sep-2015. A total of 295 participants were enrolled and randomly assigned to study treatment; 278 participants completed the study. Of the 295 participants, 167 participants were reported with Ascaris lumbricoides infestation and 243 participants were reported with Trichuris trichiura infestation.
Pre-assignment Details: Of the 792 participants screened, a total of 295 were randomly assigned to study treatments, of which 278 completed the study. 17 participants were withdrawn from study with following reasons: Withdrawal by participant (12), Lost to follow-up (3), Physician decision (1) and Protocol violation (1).
Groups:
- Double-blind Placebo: Placebo Comparator: Placebo. Matching placebo was administered as a single-dose chewable tablet in a double-blind manner at the baseline visit (Day 1) followed up to Visit 3 (Day 19+/-2).
- Double-blind Mebendazole 500 mg: Experimental: Mebendazole. Mebendazole was administered as a single 500-mg chewable tablet in a double-blind manner at the baseline visit (Day 1) followed up to Visit 3 (Day 19+/-2).
- Open-label Mebendazole 500 mg: Mebendazole 500-mg chewable tablet was administered in an open label manner at visit 3 (Day 19+/-2) followed up to Visit 5 (Day 7+/-1 from Visit 3).
Period: Double-blind
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg | Open-label Mebendazole 500 mg
Started | 146 | 149 | 0
Completed | 137 | 141 | 0
Not Completed | 9 | 8 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7 | 0
Period: Open-label
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg | Open-label Mebendazole 500 mg
Started | 0 | 0 | 278
Completed | 0 | 0 | 278
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg | Total
Number analyzed (Participants) | 146 | 149 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (3.09) | 7.9 (3.27) | 7.8 (3.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 152
  Male | 72 | 71 | 143
Region of Enrollment [Number; unit: participants]
  ETHIOPIA | 127 | 128 | 255
  RWANDA | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate for Ascaris Lumbricoides at the End of Double-blind Treatment Period
Description: Cure is defined as a post-treatment egg count of zero in participants who had a positive egg count at baseline.
Time Frame: At Visit 3 (Day 19) of Double-blind treatment period
Population: The intent-to-treat (ITT) analysis set included all randomized participants with a pretreatment stool sample positive for 1 or more worms of interest. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg
Number analyzed (Participants) | 81 | 86
percentage of participants | 11.1 [5.2 to 20.1] | 83.7 [74.2 to 90.8]
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Mebendazole 500 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Cure Rate for Trichuris Trichiura at the End of Double-blind Treatment Period
Description: Cure is defined as a post-treatment egg count of zero in participants who had a positive egg count at baseline.
Time Frame: At Visit 3 (Day 19) of Double-blind treatment period
Population: The ITT analysis set included all randomized participants with a pretreatment stool sample positive for 1 or more worms of interest. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg
Number analyzed (Participants) | 119 | 124
percentage of participants | 7.6 [3.5 to 13.9] | 33.9 [25.6 to 42.9]
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Mebendazole 500 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Event (TEAE) in Double-Blind Treatment Period
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to Visit 3 (Day 19 +/-2)
Population: The safety analysis set consisted of all randomized participants who received 1 dose of study agent (mebendazole or placebo) at baseline. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg
Number analyzed (Participants) | 140 | 144
participants | 8 | 9

4. Secondary Outcome: Egg Count Reduction Rate (Percent) for Ascaris Lumbricoides Infestation at the End of Double-blind Treatment Period
Description: Percent egg count reduction is calculated as average egg count at end of treatment period of a treatment group minus average egg count at baseline of the treatment group divided by average egg count at baseline of the treatment group.
Time Frame: Baseline and Day 19 (Visit 3) at the End of Double-blind Treatment Period
Population: as for outcome 2
Measure: Number; unit: percent change in egg count
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg
Number analyzed (Participants) | 81 | 86
percent change in egg count | -19.2 (20684.03) | -97.9 (23476.82)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Mebendazole 500 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Egg Count Reduction Rate (Percent) for Trichuris Trichiura Infestation at the End of Double-blind Treatment Period
Description: as for outcome 4
Time Frame: Baseline and Day 19 (Visit 3) at the End of Double-blind Treatment Period
Population: as for outcome 2
Measure: Number; unit: percent change in egg count
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg
Number analyzed (Participants) | 119 | 124
percent change in egg count | -10.5 (930.05) | -59.7 (1256.22)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Mebendazole 500 mg; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Mebendazole
Description: The Cmax is the maximum plasma concentration.
Time Frame: Predose, 1, 2, 3, 5, 8 and 24 hours postdose at visit 4 (Day 20; 1 day after Visit 3)
Population: Pharmacokinetic (PK) population included all randomized participants who received at least 1 dose of the study drug and had valid pharmacokinetic profile. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per Milliliters (ng/mL)
Groups:
- Mebendazole: Group 1 (1 to <3 Years): Group 1 represents pharmacokinetic analysis set which included participants with age group 1 to less than (<) 3 years and received Mebendazole 500 milligram (mg).
- Mebendazole: Group 2 (3 to 6 Years): Group 2 represents pharmacokinetic analysis set which included participants with age group 3 to 6 years and received Mebendazole 500 mg.
- Mebendazole: Group 3 (7 to 16 Years): Group 3 represents pharmacokinetic analysis set which included participants with age group 7 to 16 years and received Mebendazole 500 mg.
Arm/Group | Mebendazole: Group 1 (1 to <3 Years) | Mebendazole: Group 2 (3 to 6 Years) | Mebendazole: Group 3 (7 to 16 Years)
Number analyzed (Participants) | 22 | 12 | 10
nanogram per Milliliters (ng/mL) | 210.0 (212.0) | 49.9 (26.8) | 34.2 (13.8)

7. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Event (TEAE) in Open-Label Treatment Period
Description: as for outcome 3
Time Frame: At Visit 3 (Day 19+/-2) followed up to Visit 5 (Day 7+/-1 from Visit 3)
Population: The open-label follow-up safety analysis set consisted of all randomized participants who received a 500-mg chewable tablet of mebendazole at Visit 3. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Open-label Mebendazole 500 mg
Number analyzed (Participants) | 278
participants | 7

8. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Mebendazole
Description: The Time to Reach Maximum Plasma Concentration (Tmax) is time to reach the maximum plasma concentration.
Time Frame: Predose, 1, 2, 3, 5, 8 and 24 hours postdose at visit 4 (Day 20; 1 day after Visit 3)
Population: PK population included all randomized participants who received at least 1 dose of the study drug and had valid pharmacokinetic profile. Here 'N' signifies number of participants analysed for this outcome measure.
Measure: Mean (Full Range); unit: hours
Arm/Group | Mebendazole: Group 1 (1 to <3 Years) | Mebendazole: Group 2 (3 to 6 Years) | Mebendazole: Group 3 (7 to 16 Years)
Number analyzed (Participants) | 22 | 12 | 10
hours | 2.5 [1 to 8] | 2 [0.98 to 3] | 3 [1 to 8]

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours (AUC8h) of Mebendazole
Description: The (AUC8h) is the area under the plasma concentration-time curve from time 0 to 8 hours Post-dose.
Time Frame: Predose, 1, 2, 3, 5, 8 and 24 hours postdose at visit 4 (Day 20; 1 day after Visit 3)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanogram hour per Milliliters(ng*h/mL)
Arm/Group | Mebendazole: Group 1 (1 to <3 Years) | Mebendazole: Group 2 (3 to 6 Years) | Mebendazole: Group 3 (7 to 16 Years)
Number analyzed (Participants) | 21 | 9 | 10
nanogram hour per Milliliters(ng*h/mL) | 697 (367) | 242 (139) | 182 (66.3)

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-last) of Mebendazole
Description: The (AUC [0-last]) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Time Frame: Predose, 1, 2, 3, 5, 8 and 24 hours postdose at visit 4 (Day 20; 1 day after Visit 3)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Mebendazole: Group 1 (1 to <3 Years) | Mebendazole: Group 2 (3 to 6 Years) | Mebendazole: Group 3 (7 to 16 Years)
Number analyzed (Participants) | 22 | 12 | 10
ng*h/mL | 1320 (844) | 416 (215) | 387 (190)

ADVERSE EVENTS:
Time Frame: Up to visit 5 (Day 26, 7+/-1 days after Visit 3 [Day 19+/-2])
Groups:
- OL Mebendazole 500 mg: Mebendazole 500-mg chewable tablet was administered in an open label manner at visit 3 (Day 19+/-2) followed up to Visit 5 (Day 7+/-1 from Visit 3).
Arm/Group | Double-blind Placebo | Double-blind Mebendazole 500 mg | OL Mebendazole 500 mg
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/144 | 0/278
Other Adverse Events (participants affected / at risk) | 8/140 | 9/144 | 7/278
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=140) | Double-blind Mebendazole 500 mg (N=144) | OL Mebendazole 500 mg (N=278)
Night Blindness (Eye disorders) | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis Bacterial (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Tinea Infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vitamin A Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.